CLINICAL TRIAL: NCT06046768
Title: The Consequences of Child Verbal and Eating Disorders on Family Dynamics in the Context of Ear Nose and Throat (ENT) Pathologies - Integration of Non-verbal Communication and Parental Support
Brief Title: Assessment and Remediation of Oral Disorders
Acronym: ERTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230152; IDRCB: 2023-A00202-43 (Registry Identifier: ANSM)
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Oral Disorder
Keywords: parental stress; ENT pathology
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Intervention Model Description: To evaluate the impact of psychological treatment on the improvement of oral disorders perceived by parents in their child.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Child with oral feeding disorder(s) (Experimental): Child (boy or girl) with oral feeding disorder(s) diagnosed by a speech therapist as part of a speech therapy assessment.
  Interventions: Other: Psychological care

INTERVENTIONS:
Other: Psychological care — Psychological consultations (interviews, scales), participation in a discussion group for parents in Visio via Zoom, a speech therapy assessment and possible complementary multidisciplinary consultations)

SUMMARY:
As part of the Reference Center for Rare Diseases of the Robert Debré Hospital, many children have eating and verbal oral disorders. In this doctoral research, we question the psychological impact of oral disorders on the dynamics of family functioning.Our research entitled: Evaluation and Remediation of Orality Disorders (ERTO) aims to evaluate the impact of psychological care of the child and a support program for parents.

We hypothesized that this comprehensive management could contribute to improving disorders and consequently modify parental representations of the child and his disorders.

In addition, care focused on intra-family relations and communication would allow a decentralization and a repositioning of the problem of disorders within the family dynamic.

The results of this research will have concrete applications for the management of children suffering from oral disorders.

DETAILED DESCRIPTION:
The ERTO search follows the first PREORA search. As soon as the results of the PREORA questionnaires are obtained, we would constitute a cohort of 16 children - a maximum of 32 parents and siblings. It will be extracted from participants in the PREORA study by random draw after screening eligibility according to the inclusion criteria and their desire to participate in this study.

We will study a population of children aged 18 months to 3 years, with ENT pathology, requiring surgery and invasive care.

The research consists of three stages:

T0: An inclusion interview: standardized psychological interview (recorded Stern R interview and PSI Parental Stress Scale). ""R interview"" is a questionnaire published and validated in 1989 by Stern, Robert-Tissot, Besson, et al.

It allows the evaluation of maternal representations. The Parental Stress Index (PSI), translated in Quebec by Bigras and Lafrenière, is used to detect difficulties in parent-child dyads.

T1-T5: Then a follow-up will be proposed (five psychological consultations (interviews, scales), participation in a discussion group for parents in Visio via Zoom, a speech therapy assessment and possible complementary multidisciplinary consultations) T6: Again an assessment with the T0 retest (Stern R Interview, PSI Parental Stress Scale, MCH scale). This study is a non-randomized exploratory research with two controlled groups, before/after.

Parental stress and child representation will be assessed according to the two subgroups of belonging, group A (antenatal diagnosis), group B (postnatal diagnosis), t1 (before psychological management), t2 (after 5 months of psychological management) and t3 (after one year of discussion group). Qualitative and quantitative analyses will be provided, based on variables.

ELIGIBILITY:
Inclusion Criteria:

* Child (boy or girl) with oral feeding disorder(s) diagnosed by a speech therapist as part of a speech therapy assessment
* Patients under ENT care at Robert Debré Hospital
* Children aged 18 months to 3 years
* French-speaking parents
* Living at home in France
* Affiliation with a social security scheme or entitled beneficiary
* Informed consent signed by both parents

Exclusion Criteria:

* Pathologies predominantly associated with ENT pathology
* Neurological disorders
* Deafness

Ages: 18 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Parental stress and child representation | 12 months
  Montreal children's Hospital scale. Parental stress and child representation will be assessed by three times t1 (before psychological management), t2 (after 5 months of psychological management) and t3 (after one year of discussion group).

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided